CLINICAL TRIAL: NCT07361770
Title: Comparative Effect of Instrument Assisted Soft Tissue Mobilization and Cross Fiber Massage in Patients With Total Knee Replacement.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rashid Latif Medical College (Other)
Responsible Party: Principal Investigator, Kainat Zahara, House officer Physical Therapy, Rashid Latif Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB/2024/168
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Total Knee Replacement
Keywords: Instrument Assisted Soft Tissue Mobilization; Cross Fibre Massage; Pain; Range of motion; Total Knee Replacement
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Group A: IASTM Patients received IASTM with baseline treatment. Group B: Cross Fiber Massage Patients received Cross fiber massage with baseline treatment.
Who Masked: Outcomes Assessor
Masking Description: The assessor was kept blind and was not aware of any intervention groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instrument Assisted Soft Tissue Mobilization (Experimental): The Graston Technique of Soft-Tissue Therapy (GT), also known as instrument-assisted soft tissue mobilization (IASTM), is used by chiropractors, physicians, and therapists to manage pain and range-of-motion limitations caused by scar tissue and musculoskeletal injuries. The GT treats tissue injuries and pain by separating scar tissue and producing heat, which increases blood flow to the areas affected by pain or trauma.
  Interventions: Other: Instrument-assisted soft tissue mobilization
- Cross Fibre Massage (Active Comparator): Deep tissue massage is a type of massage that focuses on the muscular tissue's most profound levels. In tight regions, therapists utilize a combination of gentle strokes and deep pressure with their fingers, palms, and forearms. Either following or by going over the muscle fibers. It is used for back pain Reduce high blood pressure, Relieve pain and stiffness Speed up the healing of muscle strains and sprains Chronic constipation.
  Interventions: Other: Cross Fibre Massage

INTERVENTIONS:
Other: Instrument-assisted soft tissue mobilization — Each treatment session was of 15-20 minutes for all muscles, with the help of IASTM device assisted by friction-free oil or gel. The general principle is a six-step technique comprising examination, warm-up, IASTM, stretching, strengthening and icing. Data was collected by an independent assessor at baseline and after 4 weeks
  Arms: Instrument Assisted Soft Tissue Mobilization
Other: Cross Fibre Massage — The massage is deep and must be applied transversely to the specific tissue involved unlike the superficial massage given in the longitudinal direction parallel to the vessels which enhances circulation and return of fluid. The therapist's fingers and patient's skin must move as one, otherwise moving subcutaneous fascia against muscle or ligament could lead to blister formation or subcutaneous bruising.
  Data was collected by an independent assessor at baseline and after 4 weeks.
  Arms: Cross Fibre Massage

SUMMARY:
Comparative effect of Instrument Assisted Soft Tissue Mobilization and Cross Fiber Massage in patients with Total Knee Replacement

DETAILED DESCRIPTION:
Total knee replacement (TKR) is an elective procedure in which the knee joint is resurfaced with a metal or plastic implant intended to restore function, provide pain relief, and improve quality of life.IASTM helps to remove the scarring and decrease the pain caused by muscular tightness. The therapeutic benefits of the application of IASTM occur in a short period, including improvement in range of motion, reduction of pain, decreasing hypertonia.Cross fiber massage, is a form of massage technique that focuses on the body's deep tissues. The massage is deep and should be delivered in transverse direction to the particular tissue affected, as opposed to superficial massage applied longitudinally parallel to the vessels, which promotes circulation and fluid return.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female of Age 40-60
* Radiological diagnosis
* Advanced degenerative OA knee, undergoing a primary TKR
* Pain intensity >3

Exclusion Criteria:

* Rheumatoid Arthritis patients
* Septic Arthritis and other inflammatory arthritis patients
* Secondary or traumatic O.A
* Congenital bony deformities
* Flexion contracture, patellar dislocation
* Fracture or pervious osteotomy
* Neurological dysfunction

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Both male and female
Enrollment: 50 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Baseline and 4th week
  Visual Analogue Scale (VAS) is a widely used tool to measure pain intensity. The visual analog scale (VAS) for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. It was used to assess pain.

SECONDARY OUTCOMES:
Range Of Motion | Baseline and 4th week
  An inclinometer app is a tool that helps measure and track changes in joint mobility, flexibility, and range of motion. It provide objective, reliable degree measurements of knee range of motion and joint position sense error. These measurements are then compared against established normal ranges or the patient's own previous results to track progress.

OTHER OUTCOMES:
Knee Funtion | Baseline and 4th week
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a self-reported outcome measure assessing the patient's opinion about the health, symptoms, and functionality of their knee. It is a questionnaire, including 5 subscales: symptoms, pain, ADLs, sports/recreation, and quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Arif Memorial Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The data will be available on reasonable request from corresponding author.
Supporting Information: Study Protocol
Time Frame: It will available after publication of study.
Access Criteria: The researchers and other scientists , but after publication.

REFERENCES:
- [Result] Bhosale P, Kolke Pt S. Effectiveness of instrument assisted soft tissue mobilization (IASTM) and muscle energy technique (MET) on post-operative elbow stiffness: a randomized clinical trial. J Man Manip Ther. 2023 Oct;31(5):340-348. doi: 10.1080/10669817.2022.2122372. Epub 2022 Sep 28. PMID 36171728